CLINICAL TRIAL: NCT01149239
Title: The Effect of Preoperative Anxiety Level on the Induction Dose of Propofol and MAC-hour of Sevoflurane During Thyroidectomy
Brief Title: The Effect of Preoperative Anxiety Level on the Induction Dose of Propofol and Minimum Alveolar Concentration (MAC) Hour of Sevoflurane During Thyroidectomy
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Jeong-Yeon Hong / Associate Clinical Professor, Yonsei University, College of Medicine
Other Study IDs: 4-2010-0117
Record Dates: First submitted 2010-06-17; First posted 2010-06-28 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Thyroidectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is to evaluate the level of anxiety, and to check the correlation of induction dose and the amount of sevoflurane to keep anesthetic depth in in female patients undergoing thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* female patients (ASA physical status I and II) aged between 20-65 years and scheduled elective thyroidectomy

Exclusion Criteria:

* cardiovascular, renal, liver disease, or psychiatric disorder

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female patients aged between 20-65 years and scheduled elective thyroidectomy
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Yeon Hong, MD, Principal Investigator — Anesthesiology & Pain Medicine, Severance Hospital
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea